CLINICAL TRIAL: NCT06878027
Title: Analysis of Urinary Methylation Patterns Via Liquid Biopsy as a Tool for Early Diagnosis, Non-invasive Monitoring and Prediction of Recurrence Risk in Bladder Cancer
Brief Title: Analysis of Urinary Methylation Patterns Via Liquid Biopsy as an Early Diagnosis Tool
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Azienda Ospedaliera Santa Maria Degli Angeli (Other); Istituto per lo Studio, la Prevenzione e la Rete Oncologica (Other)
Responsible Party: Sponsor
Other Study IDs: RS194/IRE/24
Record Dates: First submitted 2025-02-12; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer
Keywords: methylation levels in urine samples
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — methylation levels in urine samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients suffering from bladder cancer: Patients with a proven diagnosis of muscle-infiltrating or non-muscle-infiltrating bladder cancer, having performance status (PS) 0-1.
- Healthy persons.: Healthy persons with no previous or current medical history associated with bladder cancer or diagnostic suspicion associated with cancer, to be used as a relative reference.

SUMMARY:
Multicenter, observational, prospective, biological pilot study on liquid biopsy, aimed at investigating methylation profiles in relation to the early diagnosis of bladder cancer, to validate the potential of commercially available tests (e.g. BladderCARE, Bladder EpiCheck), to apply and validate tests based on targeted multi-marker or genome wide analyzes via NGS and to identify methylation profiles as a tool to infer clinical outcome.

DETAILED DESCRIPTION:
The study has the primary objective to investigate the diagnostic capacity of methylation levels in urine samples, furthermore it has the secondary objective of applying an NGS test on the urine sample capable of evaluating the highest methylation levels comprehensive, with better analytical performance than the currently available standard on the market, leveraging targeted sequencing of multiple genes or global analysis of the whole methylome.

To describe the diagnostic performance of the methods in a real-world clinical environment and identify the characteristic methylation profiles capable of stratifying patients with different prognoses, and finally to explore the potential economic impact of applying such tests as tools alternatives to conventional practices.

ELIGIBILITY:
Inclusion Criteria:

Patient group

* age ≥ 18 years
* proven diagnosis of bladder cancer (infiltrating muscle or non-infiltrating muscle)
* performance status (PS) 0-1
* ability to follow the procedures established by the study
* written consent for participation in the study and data processing

group of healthy subjects

* age ≥ 18 years
* ability to follow the procedures established by the study
* written consent for participation in the study and data processing

Exclusion Criteria:

Patient group

* presence of metastatic bladder cancer
* lack of autonomy in following the procedures established by the study

group of healthy subjects

* previous or current clinical history associated with bladder cancer
* diagnostic suspicion associated with tumor pathologies
* ongoing or previous systemic oncological treatments
* presence of inflammatory and/or autoimmune diseases related to particular conditions potentially modifying the methylation profile
* existing pharmacological treatments (and/or any other type of treatment) that could alter the results of the analyzes conducted for the present study
* lack of autonomy in following the procedures established by the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by non-muscle infiltrating bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
Methylation state | 18 months
  Measurement of methylation status using the Bladder CARE test (Pangea Laboratory LLC). The test, based on quantitative PCR and evaluation of methylation status in 3 target genes, is performed on a urine sample and has reported high sensitivity (94%) and specificity (93%) values in determining the presence of bladder cancer

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Cancer Institute "Regina Elena", Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided